CLINICAL TRIAL: NCT05553275
Title: Permissive Intrapartum Glucose Control: An Equivalence Randomized Control Study (PERMIT)
Brief Title: Permissive Intrapartum Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ghamar Bitar, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0577
Record Dates: First submitted 2022-09-09; First posted 2022-09-23 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Gestational Diabetes; Pregestational Diabetes
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1:Usual Care (Active Comparator)
  Interventions: Procedure: Usual Care
- Group 2: Permissive Care (Experimental)
  Interventions: Procedure: Permissive intrapartum glucose control

INTERVENTIONS:
Procedure: Usual Care — Blood sugar evaluation (accuchecks) every four hours in latent labor and every 2 hours in active labor.Participants will be routinely managed with maintenance fluids of lactated ringers during latent labor and lactated ringers with dextrose 5% in active labor. Blood sugars of more than 110 mg/dl at any time point in labor will be treated with an insulin drip as follows:
  Regular insulin (100 units) in 100cc of normal saline, with Lactated Ringers with 5% dextrose at 125cc/hour. If blood sugar 111-140, insulin drip at 1 unit/hour will be given and continued if blood sugar is 111-140.If blood sugar is 141-180, then drip will be changed to to 1.5 unit/hour and if blood sugar is 181-220, drip will be changed to 2.0 units/hour and MD will be called if blood sugar is more than 221 mg/dl
  Arms: Group 1:Usual Care
Procedure: Permissive intrapartum glucose control — Blood sugar evaluation (accuchecks) every four hours in latent labor and every 2 hours in active labor.Participants will be routinely management with maintenance fluids of lactated ringers during latent labor and lactated ringers with dextrose 5% in active labor.Blood sugars of more than 180 mg/dl at any time point in labor will be treated with an insulin drip as follows:
  Regular insulin (100 units) in 100cc of normal saline, with Lactated Ringers with 5% dextrose at 125cc/hour.If blood sugar is 181-200, insulin drip at 1 unit/hour will be given. If blood sugar is 201-220, then drip will be changed to 1.5 units/hour. If blood sugar is 221 - 250, then drip will be changed to 2.0 units/hour and if blood sugar is more than 251 MD will be called.
  Arms: Group 2: Permissive Care

SUMMARY:
The purpose of this study is to assess whether permissive intrapartum glycemic control compared to usual care would lead to similar rate of neonatal hypoglycemia among people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Presenting for intrapartum management (induction, labor, augmentation)
* Any diagnosis of Type 1 Diabetes Mellitus(T1DM), Type 2 Diabetes Mellitus (T2DM), or Gestational Diabetes
* English or Spanish fluency

Exclusion Criteria:

* Major fetal anomalies affecting glucose metabolism
* Multiple Gestation
* Incarcerated subjects
* less than 34 weeks gestation of pregnancy
* Planned cesarean delivery
* Utilizing insulin pump during labor
* Stillbirth
* Presenting in Diabetic ketoacidosis(DKA)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
first neonatal blood glucose level measured in mg/dL | up to 2 hours of life prior to first feed

SECONDARY OUTCOMES:
Number of intrapartum glucose measurements | During Labor(for up to 200 hours)
Mean maternal glucose values in mg/dl | during latent labor(for up to 200 hours)
Mean maternal glucose values in mg/dl | during active labor(for up to 200 hours)
Overall mean maternal glucose values in mg/dl | in all of labor(for up to 200 hours)
Number of participants that have hyperglycemia episodes | during labor( for up to 200 hours)
  Hyperglycemia is defined as blood sugar levels greater than 200 mg/dl
Number of participants that have hypoglycemia episodes | during labor(for up to 200 hours)
  Hypoglycemia is defined as blood sugar levels less than or equal to 60 mg/dl or symptomatic or requiring IV dextrose
Number of participants that have Diabetic Ketoacidosis | during labor(for up to 200 hours)
  Diabetic Ketoacidosis includes uncontrolled hyperglycemia, anion gap metabolic acidosis, and ketosis
Maximum insulin Glucose tolerance test (GTT) rate | during labor(for up to 200 hours)
Number of participants that utilize insulin drip | during labor(for up to 200 hours)
Number of participants that undergo primary cesarean section | at time of delivery
Number of participants that have Postpartum hemorrhage | from discharge until 6 months after birth
  Postpartum hemorrhage is defined as greater than or equal to 1000ml or need for blood transfusion
Number pf participants that have Intra-amniotic Infection | intrapartum or within 24 hours of delivery
  Intra-amniotic Infection is defined as clinically diagnosed infection of the uterine environment
Number pf participants that have endometriosis | Between 24 hours after delivery to 6 weeks of delivery
  Endometritis is defined as clinically diagnosed uterine infection
Number pf participants that have wound complications | within 6 weeks of delivery
  Wound complications is defined as superficial or deep infections, fascial dehiscence
Number pf participants that require blood product transfusion | during admission (for up to 6 weeks after neonate delivery)
Resource utilization during labor as assessed by the number of accuchecks done | during delivery admission (labor or induction/augmentation) until delivery defined as time patient is admitted to labor and delivery until birth time of neonate, for up to 200 hours
Resource utilization during labor as assessed by the number of nurses utilized | during delivery admission (labor or induction/augmentation) until delivery defined as time patient is admitted to labor and delivery until birth time of neonate, for up to 200 hours
Total facility and physician costs for all the services provided to the mothers | From maternal admission time to maternal discharge time(upto 6 months form admission date)
Total facility and physician costs for all the services provided to the neonates | from birth time to discharge time defined as birth time of neonate until neonate is discharged from the hospital, up to 1 year
Total nurse time cost for monitoring the patients during labor | From admission time to delivery time defined as time patient is admitted to labor and delivery until birth time of neonate, for up to 200 hours
Number of gestational diabetes participants that do an oral glucose tolerance test (OGTT) | within 6- 8 weeks of delivery
Neonatal C-peptide levels from cord blood | at time of delivery
Number of neonates that have blood glucose level less than 40 mg/dL | within the first 24 hours of life
Number of neonates that have blood glucose level less than 40 mg/dL | during birth admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Number of neonates that need oral glucose supplementation | during birth admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Number of neonates that need IV glucose | during birth admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Lowest neonatal glucose level | during birth admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Mean neonatal glucose level in first 24 hours of life | during birth admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Lowest neonatal glucose level | first 24 hours of life
Number of neonates that required shoulder dystocia | at time of delivery
  Shoulder dystocia is defined as the need for any extra maneuvers, other than gentle downward traction of the fetal head to deliver the fetal body after the fetal head has been delivered
Number of neonates that had birth injury | from birth and during admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
  Birth injury as defined as skull, clavicular, humerus fracture, or brachial plexus
Number of neonates that had respiratory distress | first 24 hours of life
  Respiratory distress is defined as the need for at least 4 hours of respiratory support with supplemental oxygen, continuous positive airway pressure, or ventilation
Number of fetal deaths | during labor defined as time patient is admitted to labor and delivery until birth time of neonate, for up to 200 hours
Number of neonatal deaths | within 28 days of birth
Number of neonates with Apgar score of less than 7 | 5 minutes from birth
Number of neonates that are admitted to Neonatal intensive care unit (NICU) | from birth up to 6 months from birth
Number of days neonates are admitted to NICU | from birth up to 6 months from birth
Number of neonates that have neonatal hyperbilirubinemia requiring phototherapy | during admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Maximum Bilirubin level | during admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Number of neonates that have hypocalcemia | during admission defined as birth time of neonate until neonate is discharged from hospital, up to 1 year
Number of neonates that have Necrotizing Enterocolitis | from birth up to 6 months from birth
Number of neonates that are small for gestational age | at birth
  Small for gestational age is defined as a weight below 10th percentile of the expected value according to gestational age
Number of neonates that are large for gestational age | at birth
  Large for gestational age is defined as a weight above 90th percentile of the expected value according to gestational age
Number of neonates that have Macrosomia | at time of birth
  Macrosomia is defined as weight more than 4000 grams

CONTACTS AND LOCATIONS:
Overall Officials: Ghamar Bitar, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Michal F Bartar, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No